CLINICAL TRIAL: NCT02058251
Title: Oxytocin Suppresses Substance Use Disorders Associated With Chronic Stress
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 018127-002 Seq. 1
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-12

CONDITIONS: Alcohol Use Disorders
Keywords: Alcohol; Oxytocin; Stress reactivity
MeSH Terms: conditions — Alcoholism | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): Each participant will self-administer a 40 IU dose of intranasal oxytocin.
  Interventions: Drug: Oxytocin
- Control (Placebo Comparator): Each participant will self-administer a 40 IU dose of intranasal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — One 40 IU dose of intranasal oxytocin will be self-administered (5 puffs in each nostril) by participants.
  Arms: Oxytocin
Drug: Placebo — Each participant will self-administer a 40 IU dose of intranasal saline.
  Arms: Control

SUMMARY:
In comparison to the general population, military personnel and veterans are at increased risk of developing both substance use disorders (SUDs) and post-traumatic stress disorder (PTSD). Despite promising developments in the past decade, the treatment of patients with SUDs and comorbid PTSD is woefully inadequate (Back, 2010; Back et al., 2014; Brady et al., 2007; McCauley et al., 2012). One of the adverse effects of abused drugs is their long-term negative impact on social behavior that is thought to involve oxytocin (OT) dysregulation (McGregor et al., 2008). In preclinical and clinical experiments, local, intra-nasal, or systemic OT administration decreases activation of the amygdala in response to visual fearful/threatening stimuli (Kirsch et al., 2005), ameliorates the effects of stressful events, and decreases drug-taking and seeking behavior (McGregor et al., 2008; Baskerville and Douglas, 2010; Carson et al., 2010a; Bowen et al., 2011; Cox et al 2013). However, little attention has been focused on whether OT decreases SUD vulnerability after exposure to traumatic stress in preclinical or clinical studies. This clinical project will determine whether intra-nasally administered OT will decrease craving (Aim 1) to use alcohol and decrease stress reactivity (Aim 2) following exposure to laboratory-induced stress (Trier Social Stress Task) among veterans with a dual diagnosis of alcohol use disorder and PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; any race or ethnicity; age 21-65 years.
* Female subjects will be required to complete the laboratory testing during the early to mid-follicular phase of their menstrual cycle (days 1-7 following the onset of menses).
* Veteran of the US military; any service branch.
* Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of the assessment instruments.
* Subjects must be able to comprehend English.
* Meet DSM-5 criteria for a current alcohol use disorder (assessed via the Mini International Neuropsychiatric Interview; MINI). Note that we will use the currently available diagnostic measure (MINI for DSM-IV) and will make appropriate modifications to update for compatibility with DSM-5.
* Meet DSM-5 criteria for current PTSD (assessed via the Clinician Administered PTSD Scale; CAPS). Note that we will use the currently available assessment instrument (CAPS for DSM-IV), and will make appropriate modifications to update for compatibility with DSM-5.
* A CAPS score of 50 or greater.
* Subjects will be required to have at least 5 days of abstinence from alcohol or other substances (except caffeine or nicotine) prior to completing the laboratory testing, as verified by multiple methods including self-report, breathalyzer tests, and urine drug screen tests.
* Subjects may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or anxiety disorders (e.g., agoraphobia, social phobia, generalized anxiety disorder). The inclusion of subjects with affective and anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with PTSD and alcohol use disorders.
* Subjects taking psychotropic medications will be required to be maintained on a stable dose for at least eight weeks before study initiation. This is because initiation or change of psychotropic medications during the course of the trial may interfere with interpretation of results.
* Must consent to random assignment to oxytocin or placebo.

Exclusion Criteria:

* Subjects meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders, or with current suicidal or homicidal ideation and intent. Those subjects will be referred clinically.
* Subjects who would present a serious suicide risk or who are likely to require hospitalization during the course of the study. Those subjects will be referred clinically.
* Subjects on maintenance anxiolytic, antidepressant, or mood stabilizing medications, which have been initiated during the past 8 weeks.
* Subjects with a history of a major medical illness (e.g., endocrine, cardiovascular, central nervous system disorders, peripheral neuropathy, or pulmonary disease) or other acute or unstable medical condition that might interfere with safe conduct of the study or accurate interpretation of the results.
* Subjects meeting DSM-5 criteria for another substance use disorder, except caffeine or nicotine, within the past 12 months.
* Subjects experiencing withdrawal symptoms, as evidence by a score of 10 or above on the Clinical Institute Withdrawal Assessment of Alcohol (CIWA)
* Females who are unable or unwilling to be scheduled for lab testing during the early to mid-follicular phase of their menstrual cycle.
* Pregnant women will be excluded from the proposed study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudie E. Back, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Melkonian AJ, Flanagan JC, Calhoun CD, Hogan JN, Back SE. Craving Moderates the Effects of Intranasal Oxytocin on Anger in Response to Social Stress Among Veterans With Co-Occurring Posttraumatic Stress Disorder and Alcohol Use Disorder. J Clin Psychopharmacol. 2021 Jul-Aug 01;41(4):465-469. doi: 10.1097/JCP.0000000000001434. PMID 34121063
- [Derived] Flanagan JC, Allan NP, Calhoun CD, Badour CL, Moran-Santa Maria M, Brady KT, Back SE. Effects of oxytocin on stress reactivity and craving in veterans with co-occurring PTSD and alcohol use disorder. Exp Clin Psychopharmacol. 2019 Feb;27(1):45-54. doi: 10.1037/pha0000232. Epub 2018 Nov 1. PMID 30382728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Control
Started | 35 | 38
Completed | 35 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Control | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.94 (9.75) | 47.82 (11.27) | 48.36 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 32 | 35 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 19 | 44
  White | 8 | 18 | 26
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving
Description: Using the Visual Analogue Scale (VAS), participants provided self-report ratings of subjective alcohol cravings on a scale of 1-10, with one being the lowest/better score, and 10 being the highest/worst outcome.
Time Frame: 2 hours
Population: Main outcomes analyses were limited to male participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin | Control
Number analyzed (Participants) | 32 | 35
scores on a scale | 2.89 (2.63) | 3.08 (2.71)

2. Secondary Outcome: Stress Reactivity
Description: Salivary Cortisol (μg/dL). Greater cortisol levels are indicative of greater stress reactivity.
Time Frame: 2 hours
Population: Main outcomes analyses were limited to male participants.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Oxytocin | Control
Number analyzed (Participants) | 32 | 35
μg/dL | .14 (.10) | .10 (.10)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Oxytocin | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 0/35 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No